CLINICAL TRIAL: NCT02700763
Title: PET Imaging of [18F]Dabrafenib Distribution and Kinetics in Brain Metastasis in Patients With BRAF Positive Metastastic Melanoma. A Feasibility Study.
Brief Title: [18F]Dabrafenib Molecular Imaging in Melanoma Brain Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the very low inlcusion rate and the current COVID-19 pandemic.
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201600134
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma
Keywords: Brain metastasis
MeSH Terms: conditions — Melanoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]dabrafenib molecular imaging (Experimental): A [18F]dabrafenib PET scan will be performed at baseline (7 days or less before the start of treatment with oral dabrafenib).
  Interventions: Other: [18F]dabrafenib molecular imaging

INTERVENTIONS:
Other: [18F]dabrafenib molecular imaging — A [18F]dabrafenib dynamic PET scan of the brain (60 minutes) and static total body PET scan will be performed at baseline.

SUMMARY:
In this feasibility study, [18F]dabrafenib will be used as radioactive tracer. All patients in this study are diagnosed with advanced melanoma with evidence of brain metastases and are eligible for treatment with dabrafenib, a specific V600-mutated BRAF inhibitor. Patients will undergo a dynamic PET scan of the brain to determine [18F]dabrafenib distribution and kinetics in brain metastases. In addition, a static total body PET scan will be performed to visualize whole body distribution and tracer uptake.

DETAILED DESCRIPTION:
Rationale: Dabrafenib is an oral protein tyrosine kinase inhibitor which specifically targets mutated BRAF protein. It is used in the treatment of metastatic melanoma with evidence of a BRAF V600 mutation in genomic material. However, in this group of patients often a heterogenic response to treatment is seen. Heterogeneity in drug accumulation in the tumor could be responsible for the observed differences in treatment response between lesions and between patients. Besides poor tumor accumulation of the drug, heterogeneous expression of the drug target, B-Raf protein, between patients and between lesions within a single patient could account for heterogeneity in treatment response.

PET imaging with radioactively labeled carrier-added [18F]dabrafenib (low specific activity) as the tracer might be a useful tool to show the distribution pattern and kinetics of the native drug; in particular PET can be used to determine if dabrafenib can cross the blood-brain barrier (BBB) and accumulate in brain metastases.

Since the behavior of [18F]dabrafenib in patients is hitherto unknown, first a feasibility study is needed. In this feasibility study, we will use low specific activity [18F]dabrafenib, for which a labeling procedure has already been developed, to determine the whole body distribution and kinetics in brain metastases in metastatic BRAF V600 mutation positive melanoma patients.

Study design: This study is a feasibility study for the use of [18F]dabrafenib as a PET tracer, in 10 patients. Patients who will be eligible for this study are at least 18 years of age. They are all diagnosed with metastatic melanoma with presence of metastasis to the brain and should have a positive BRAF V600 mutation status. In addition, patients should be naïve to treatment with a BRAF or MEK inhibitor.

Interventions: A [18F]dabrafenib PET/CT scan and an MRI scan of the brain will be performed at baseline, 7 days or less before the start of treatment with oral dabrafenib. CT and MRI are part of the regular care. The PET procedure commence with the injection of approximately 200 MBq [18F]dabrafenib, which is followed by a 60 minutes dynamic PET scan of the brain and thereafter a total-body PET scan (toe to head). During the dynamic PET scan of the brain, arterial blood sampling and analysis of plasma metabolites will be performed. Treatment response will be monitored as part of the regular treatment (CT for thorax/abdomen and MRI for brain) after 4 weeks. In addition, a single venous blood sample will be collected for isolation of circulating tumor DNA. Immunohistochemical staining for mutated B-raf protein will be performed on tumor tissue, either derived from a fresh biopsy or from a preexisting tumor specimen.

Nature and extent of burden and risk associated with participation, benefit and group relatedness: Patients who will participate in this study will receive a dynamic PET/CT scan of the brain, a static total-body PET/CT scan and an MRI scan of the brain at baseline. After 4 weeks they receive a CT scan of chest and abdomen and a MRI scan of the brain. All CT and MRI scans are part of regular care. The PET/CT scan, which is a study procedure, carries a radiation burden of 4.1 mSv. This constitutes an intermediate risk, based on criteria of the International Commission on Radiological Protection. For the purpose of pharmacokinetic modeling, an arterial catheter will be placed which is an invasive procedure. Expected adverse events will be identical to that of unlabeled dabrafenib. Patients do not directly benefit from the study, but their participation helps to get more insights in the pharmacokinetics of dabrafenib and its role in the treatment of brain metastases.

ELIGIBILITY:
Inclusion criteria:

1. Has signed informed consent.
2. Age >=18 years of age.
3. Histologically confirmed cutaneous metastatic melanoma (Stage IV), including confirmed brain metastases.
4. BRAF mutation-positive (V600 E/K) melanoma as determined by standardized genetic testing.
5. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. Eligible for treatment with dabrafenib. Specific information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the study treatment that may impact subject eligibility is provided in the summary of product characteristics (SPC) for Tafinlar.
7. No contraindication for performing a CT scan.
8. No contraindications for performing an MRI scan of the brain.
9. Able to swallow and retain oral medication.
10. Women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control, as defined in Section 5.2, from 14 days prior to randomization, throughout the treatment period and for 4 weeks after the last dose of study treatment.
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
12. Must have adequate organ function as defined in Table 1. Table 1 Definitions for Adequate Baseline Organ Function System Laboratory Values Hematologic ANC >= 1.2 × 109/L Hemoglobin >= 9 g/dL Platelet count >= 75 x 109/L PT/INRa and PTT <= 1.3 x ULN Hepatic Total bilirubin <= 1.5 x ULN AST and ALT <= 2.5 x ULN Renal Serum creatininec <= 1.5 mg/dL Cardial ECG QTc < 480 msec Abbreviations: ALT = alanine transaminase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ECG = electrocardiogram; INR = international normalized ratio; PT = prothrombin time; PTT = partial thromboplastin time; ULN = upper limit of normal.

    1. Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to randomization.
    2. Except subjects with known Gilbert's syndrome.
    3. If serum creatinine is > 1.5 mg/dL, calculate creatinine clearance using standard Cockcroft-Gault formula. Creatinine clearance must be >= 50 mL/min to be eligible.
13. Women of child-bearing potential must have a negative urine or serum pregnancy test (β-HCG) within 14 days of first dose of study treatment.

Exclusion Criteria:

1. Previous treatment with a BRAF or MEK inhibitor. (previous systemic treatment for melanoma with other agents is allowed).
2. Previous brain surgery or radiotherapy to the brain.
3. Cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, vaccine therapy or major surgery) or investigational anti-cancer drugs within the last 3 weeks, or chemotherapy without delayed toxicity within the last 2 weeks, preceding the first dose of dabrafenib.
4. Current use of a prohibited medication or requires any of these medications during treatment with dabrafenib as mentioned in the SPC for Tafinlar.
5. Current use of oral anticoagulant therapy. NOTE: Prophylactic low-dose of low molecular weight heparin (LMWH) is permitted.
6. Known immediate or delayed hypersensitivity reaction to dabrafenib or excipients.
7. Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study treatment and during the study.
8. Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (26) grade 2 or higher from previous anti-cancer therapy, except alopecia.
9. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, the Novartis medical monitor will be contacted.
10. Presence of malignancy other than disease under study within 5 years of study enrollment, or any malignancy with confirmed activating RAS mutation. Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
11. Leptomeningeal metastases, brain metastases, or metastases causing spinal cord compression that are symptomatic or not stable for >=4 weeks or requiring corticosteroids. Subjects on a stable dose of corticosteroids >1 month or who have been off of corticosteroids for at least 2 weeks can be enrolled with approval of the Novartis medical monitor.
12. A history or evidence of cardiovascular risk including any of the following:

    1. A QT interval corrected for heart rate using the Bazett's formula >=480 msec;
    2. A history or evidence of current clinically significant uncontrolled arrhythmias;
    3. A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
    4. A history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines.
    5. Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
    6. Patients with intra-cardiac defibrillators.
13. A history of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and/or HCV will be permitted).
14. Any serious or unstable pre-existing medical conditions (i.e, diabetes mellitus, hypertension, etc), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
15. Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent, unless a legally acceptable representative could provide informed consent.
16. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Absolute uptake of [18F]dabrafenib | 60 minutes
  Determination of the absolute uptake (Standard uptake value (SUV)) and kinetics (time-activity curves, volume of distribution) of [18F]dabrafenib in normal brain and brain metastasis.

SECONDARY OUTCOMES:
Heterogeneity of [18F]dabrafenib uptake of tumor lesions and kinetics in the brain | Baseline
  Analysis of heterogeneity in [18F]dabrafenib accumulation and kinetics between lesions within one organ (brain; intra-patient heterogeneity).
Intra-patient heterogeneity in [18F]dabrafenib uptake of tumor lesions | Baseline
  Analysis of heterogeneity in [18F]dabrafenib accumulation between lesions in different organs including brain metastases (total body imaging; intra-patient heterogeneity).
Inter-patient heterogeneity in [18F]dabrafenib uptake of tumor lesions | baseline
  Analysis of heterogeneity in [18F]dabrafenib accumulation between all lesions in different patients (Inter-patient heterogeneity).
Correlation of [18F]dabrafenib uptake with response to dabrafenib treatment of tumor lesions | 4 weeks
  Correlation of accumulation of [18F]dabrafenib in melanoma metastasis with response to treatment according to the RECIST criteria (response evaluation with MRI brain and CT of chest and abdomen after 4 weeks).
Correlation between absolute tumor tracer uptake of [18F]dabrafenib and immunohistochemical staining with VE1 mAb (anti V600-mutated BRAF). | Baseline
  Correlation between absolute tumor tracer uptake of [18F]dabrafenib and positive immunohistochemical staining using specific MAB's against mutated B-Raf protein.
Correlation between absolute tumor tracer uptake of [18F]dabrafenib and BRAF V600 mutation load as maesured in circulating tumor DNA (ctDNA). | Baseline
  Correlation between absolute tumor tracer uptake of [18F]dabrafenib and BRAF V600 mutation load in ctDNA as measured by quantitative PCR.
Comparison between direct DNA sequencing and Droplet Digital Polymerase Chain Reaction (ddPCR) for BRAF mutation detection. | Baseline
  Correlation between BRAF mutation status as determined by direct DNA sequencing using tumor tissue samples (golden standard) and ddPCR using ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Geke AP Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No